CLINICAL TRIAL: NCT06791525
Title: Single-arm, Open-label Study of Tirbanibulin 1% Ointment to Treat Warts on the Hands in Pediatric Patients
Brief Title: Tirbanibulin for Pediatric Warts
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Skin Center Dermatology Group (Industry)
Responsible Party: Principal Investigator, Dr. Peter C. Friedman, Principal Investigator, The Skin Center Dermatology Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIRBAVV
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Warts Hand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical treatment arm (Experimental): Topical medication self-applied
  Interventions: Drug: Tirbanibulin ointment 1%

INTERVENTIONS:
Drug: Tirbanibulin ointment 1% — Topical application

SUMMARY:
Warts are common, benign skin lesions caused by the human papillomavirus (HPV). Treatment is challenging, particularly in the pediatric population, where standard modalities such as cryotherapy and intralesional immunotherapy are poorly tolerated. Existing topical treatments, such as imiquimod and 5-fluorouracil, have low efficacy and require prolonged use. Case reports suggest tirbanibulin ointment may provide an effective and well-tolerated alternative for pediatric warts. This study will evaluate the efficacy and safety of tirbanibulin ointment in treating pediatric hand warts.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-18
2. Subject and their legally authorized representative must be able to understand and be willing to adhere to all protocol requirements and voluntarily sign and date informed consent and assent for minors.
3. Subject is judged to be in good health as determined by the Principal Investigator, based upon the results of the screening assessments and medical history.
4. Diagnosis of warts on the hands
5. Wart count on the hands and 3-10

Exclusion Criteria:

1. Wart duration >2 years.
2. More than 10 warts in non-hand areas.
3. Total wart surface area on the hands bigger than 100 cm2
4. Prior treatment failure with the following modalities:

1. intralesional immunotherapy 2. intralesional bleomycin, 5-fluorouracil, methotrexate 3. intralesional cidofovir 5. Any over the counter, prescription topical, or in-office procedural wart treatment within 6 weeks of baseline (Day 1) 6. Known immuno-suppressed state due to disease or medication, medical treatment o 7. Known allergy to any component of the IP 8. Any conditions that, in the Principal Investigator's opinion, may interfere with the course of the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Resolution | 2 months aftre completion of 4 or less treatment cycles
  Ful resolution of treated lesions

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided